CLINICAL TRIAL: NCT03399916
Title: TranSITion: Ecological Momentary Determinants of Sedentary Behavior
Brief Title: Ecological Momentary Determinants of Sedentary Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: American College of Sports Medicine (Other)
Responsible Party: Principal Investigator, Matthew P Buman, PhD, Associate Professor, Arizona State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004349
Record Dates: First submitted 2017-12-22; First posted 2018-01-17 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: PART B: A three-factor design with two-levels yielded eight experimental conditions, half of which encouraged standing more (stand; n prompt types = 80, n total prompts =800) and the other half encouraged moving more (move; n prompt types = 80, n total prompts =800).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prompt (Experimental): An email based prompt was sent- containing either a stand or move message. Exploratory variations of the prompt were designed to include the addition of a goal e.g., stand for the next 5-minutes, and/or employer support e.g., PTS says "stand for the next 5 minutes".
  Interventions: Behavioral: Prompt sent
- No Prompt (No Intervention): Prompt delivery was sequentially randomized to be sent (ST) or not sent (NST) to all participants (probability of 0.5), at eight decision points per day (between 9am and 5pm), to achieve a total of 3200 randomizations across participants (160 per participant). Therefore 50% of the time, no prompt was sent.

INTERVENTIONS:
Behavioral: Prompt sent
  Arms: Prompt

SUMMARY:
A two phase trial to understand the personal, behavioral, environmental, and contextual factors that underpin sedentary behavior and to systematically test a series of contextual prompt characteristics that may lead to subsequent change in sedentary behavior.

DETAILED DESCRIPTION:
Phase 1: This is an observational study that will utilized Ecological Momentary Assessment, to determine which personal (e.g. fatigue, mood, and stress level), behavioral (e.g. watching TV, working at desk, and eating meals), environmental (e.g. being at home or work, time of the day, and weather) and contextual factors were associated with sedentary behavior. Three EMAs per day will be sent randomly sent to participants on weekdays (Monday to Friday), for four consecutive weeks (total of 20 days). During these days, participants will also wear an activPAL device to objectively measure sedentary behavior. The purpose of the study is to identify the combination of factors most likely to precede and proceed short (<30 min) and long (≥30 min) bouts of sedentary behavior.

Phase 2: A micro-randomized trial will be used to evaluate the efficacy of an email-based prompt to elicit a proximal effect (e.g., a postural response defined as a transition from seated to standing or seated to moving within 5 minutes to interrupt prolonged sitting) compared to a no prompt condition. A secondary aim of this study is to determine whether prompts that encourage standing are more likely to elicit a response than those that encourage moving. An exploratory aim is to examine whether varying the content of the stand or move prompt to include combinations of short term goals and employer approval, influence the magnitude of response.

ELIGIBILITY:
Inclusion Criteria:

* Full-time employees
* Males or females
* Ages 18-65
* Sedentary working habits (as indicated by >7 hrs/day of sedentary time at work in the Sedentary Behavior Questionnaire)
* Willing to engage in the study assessment and intervention for 10 weeks.

Exclusion Criteria:

* Non-ambulatory, pregnant
* Non-English speaking
* Diagnosis of psychiatric problems or taking psychiatric medications
* Medical history that prohibits prolonged standing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Minutes of sitting behavior (minutes/8h workday) | 40 days
  Objectively measured minutes of sitting, standardized to an 8h workday.
Minutes of standing behavior (minutes/8h workday) | 40 days
  Objectively measured minutes of standing, standardized to an 8h workday.
Minutes of light-intensity physical activity (minutes/8h workday) | 40 days
  Objectively measured minutes of light-intensity physical activity, standardized to an 8h workday.
Minutes of moderate-vigorous physical activity (minutes/8h workday) | 40 days
  Objectively measured minutes of moderate-vigorous physical activity, standardized to an 8h workday.

SECONDARY OUTCOMES:
Momentary affective state (4-item Likert Scales) | 20 days
  Affective states will be assessed using an ecological momentary survey based on the Positive and Negative Affect Scale (4-point Likert scale ranging from "not at all" to "extremely") (Range: 1-4) questionnaire. The ecological momentary assessment questions were designed to assess a range of contextual information (i.e., current office location, posture, social interaction) and physical and emotional feeling states (i.e., calmness, energy, happiness, stress, sadness, pain level, productivity, and willingness to stand/move). Each of these questions will be evaluated individually andaveraged to evaluate positive (i.e., calmness, energy, happiness) and negative (i.e., sadness and stress) affective states. An open-source app (Personal Analytic Companion App) will be used to deliver EMA questions randomly throughout a participant's workday. This will allow us to measure self-reported levels of positive or negative affect.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT03399916/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT03399916/SAP_001.pdf